CLINICAL TRIAL: NCT06640647
Title: A Randomized, Double-Blind, Dose-Escalation, Placebo-Controlled Phase Ia Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HDM1005 After a Single Subcutaneous Dose in Healthy Subjects
Brief Title: Phase Ia Clinical Study of HDM1005 Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HDM1005-101
Record Dates: First submitted 2024-05-31; First posted 2024-10-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-10

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- HDM1005 injection dose level 1 (Experimental): HDM1005 injection or placebo dose level 1 once subcutaneous injection
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 injection dose level 2 (Experimental): HDM1005 injection or placebo dose level 2 once subcutaneous injection
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 injection dose level 3 (Experimental): HDM1005 injection or placebo dose level 3 once subcutaneous injection
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 injection dose level 4 (Experimental): HDM1005 injection or placebo dose level 4 once subcutaneous injection
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 injection dose level 5 (Experimental): HDM1005 injection or placebo dose level 5 once subcutaneous injection
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 injection dose level 6 (Experimental): HDM1005 injection or placebo dose level 6 once subcutaneous injection
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 injection dose level 7 (Experimental): HDM1005 injection or placebo dose level 7 once subcutaneous injection
  Interventions: Drug: HDM1005 injection or placebo

INTERVENTIONS:
Drug: HDM1005 injection or placebo — HDM1005 injection or placebo isubcutaneous injection once

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-dose, dose-escalation Phase Ia clinical study. It is aimed to evaluate the safety, tolerability, PK and PD characteristics of HDM1005 injection in healthy adult subjects.

DETAILED DESCRIPTION:
In this study, 7 dose cohorts will be set up, with 10 subjects in each cohort, and subjects in each cohort will be randomized in a 4:1 ratio to receive HDM1005 injection or placebo via subcutaneous injection. Proposed dose cohorts include: Cohort 1 , Cohort 2 , Cohort 3 , Cohort 4, Cohort 5 , Cohort 6 , and Cohort 7. Scientific review committee (SRC) will be established to review the data in a blinded manner to confirm whether to proceed with the next cohort and determine the dose for the next cohort according to both protocol and data obtained from previous cohorts. Administration of higher dose cohorts will only be allowed when the safety and tolerability of the lower dose cohorts have been established and are acceptable. SRC composes representatives from the Sponsor (including but not limited to medical responsible, statistician, clinical pharmacologist) and investigator(s). External consultant may be invited as SRC member per specific scientific question.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese subjects aged 18 to 55 (including 18 and 55 years old), male or female subjects
2. BMI at the time of screening was between 19.0 and 32.0 kg/m2 (including 19.0 and 32.0 kg/m2), and the weight of female subjects was ≥45 kg and that of male subjects was ≥50 kg
3. Normal or abnormal vital signs, physical examination, laboratory examination, 12-lead ECG and chest imaging during the screening period have no clinical significance
4. Fertile female subjects, from 14 days before signing the ICF to 2 months after the administration of the drug, have taken and agreed to continue to take effective contraceptive measures, and have no family planning or egg donation plan; Male subjects had no plans to have children, no plans to donate sperm, and agreed to use highly effective contraceptive methods from signing ICF to 4 months after dosing
5. Be able to understand the procedures and methods of this study, voluntarily sign ICF, and be willing to strictly follow the requirements of clinical trial protocol to complete relevant procedures

Exclusion Criteria:

1. Previous diagnosis of type 1, type 2, or other types of diabetes
2. History or family history of medullary thyroid carcinoma, thyroid C-cell hyperplasia, or multiple endocrine adenomatosis type 2
3. As determined by the investigator, the subject has a co-existing disease or condition that affects gastric emptying or gastrointestinal nutrient absorption. Or a history of acute pancreatitis or acute gallbladder disease within 3 months prior to signing the ICF
4. Had any malignancy within 5 years prior to signing the ICF (except for basal cell carcinoma that has received curative treatment and is considered cured)
5. Cardiovascular and cerebrovascular diseases, gastrointestinal diseases, diabetes mellitus, medullary thyroid cancer, thyroid C cell hyperplasia, multiple endocrine adenomatosis type 2, chronic pancreatitis, and malignant tumors with obvious clinical significance were present; And any respiratory, neurological, urogenital, hematological, or endocrine disorders that may affect the safety of the subject or the findings of the study
6. Patients who have undergone major surgery within 3 months before signing the ICF, or who plan to undergo surgery during the study period
7. Known allergy to any component of the investigational drug or prior history of severe drug allergy
8. Drugs (including prescription drugs, over-the-counter drugs, Chinese herbs, health products, etc.) that have been used within 3 months before signing the ICF and have been determined by researchers to significantly affect body weight and blood sugar.
9. Participated in any clinical trial within 30 days prior to randomization or within 5 half-lives (whichever is older) after the last administration of the investigational drug in the clinical trial (except those who signed ICF and did not receive drug or device intervention)
10. Any of the auxiliary test indicators during the screening period meet the following criteria:

    1. Alanine aminotransferase >1.5x upper limit of normal (ULN), or ASpartate aminotransferase >1.5x ULN, alkaline phosphatase >1.5x ULN, or total bilirubin >1.5x ULN (subjects with Gilbert's syndrome can participate in this study if direct bilirubin ≤ULN);
    2. calcitonin ≥50 ng/L;
    3. Blood amylase or lipase >ULN;
    4. Thyroid stimulating hormone >6.0 mIU/L or <0.4 mIU/L;
    5. Hemoglobin a1C (HbA1c) ≥6.0%; Fasting blood glucose ≥6.1 mmol/L or < 3.9 mmol/L; Or OGTT 2 h blood glucose ≥7.8 mmol/L;
    6. eGFR < 60 mL/min/1.73m2;
    7. Male QTcF>450 ms, female QTcF>470 ms
11. People tested positive for infectious diseases 12 Habitual smokers, alcoholics and drug abusers;

13. Pregnant or lactating women 14. Blood donors within 3 months prior to randomization 15. In the Investigator's opinion, the subject is not suitable to participate in any other circumstances of the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Safety Outcomes | Signing informed until day 29
  The incidence, severity, and causality of adverse events (AE) and serious adverse events (SAEs) occurring during treatment, resulting in early termination of TEAEs, resulting in death of TEAEs; etc.

SECONDARY OUTCOMES:
PK Outcomes | 0-672 hour(s)
  PK parameters include, but are not limited to Area under the plasma concentration versus time curve (AUC)
PD Outcomes | Baseline to day 29
  Changes in body weight, body mass index (BMI), fasting glucose, fasting insulin, fasting C-peptide, blood lipids compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, Doctor, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, China